CLINICAL TRIAL: NCT05916859
Title: Effectiveness of Photodynamic Therapy Combined With Conventional Endodontic Treatment in the Disinfection of Root Canals in Patients With Apical Lesion: a Randomized Clinical Trial
Brief Title: Effectiveness of Photodynamic Therapy in the Disinfection of Root Canals in Patients With Apical Lesion
Acronym: PDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Naira Figueiredo Deana, Máster, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Folio N°062/21; DI21-0033 (Other Grant/Funding Number: Diufro)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Endodontic Treatment; Periapical Diseases
Keywords: Photodynamic Therapy; apical lesion; endodontic treatment; infra-red laser
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1. Placebo (Placebo Comparator): routine endodontic treatment will be applied and the application of laser will be simulated with the equipment, but no radiation will be emitted
  Interventions: Other: Group 1. Placebo
- Group 2. PDT 10 s (Experimental): Conventional ET + PDT. PDT will be carried out with diode laser with optical fibre coupled to the equipment (660 nm, 100 mW, 10 s). The photosensitizer used will be methylene blue.
  Interventions: Other: Group 2 PDT (10 s)
- Group 3: PDT 20 s (Experimental): Conventional ET + PDAT. PDAT will be carried out with diode laser with optical fibre coupled to the equipment (660 nm, 100 mW, 20 s). The photosensitizer used will be methylene blue.
  Interventions: Other: Group 3 PDT 20 s

INTERVENTIONS:
Other: Group 2 PDT (10 s) — - Conventional endodontic treatment associated with PDT (10 s)
  Arms: Group 2. PDT 10 s
Other: Group 3 PDT 20 s — Conventional endodontic treatment associated with PDAT (20 s)
  Arms: Group 3: PDT 20 s
Other: Group 1. Placebo — Conventional endodontic treatment
  Arms: Group 1. Placebo

SUMMARY:
The object of the present study is to compare the effectiveness of conventional endodontic treatment with that of endodontic treatment combined with Photodynamic Therapy (PDT) in patients with apical lesion. Clinical and radiographic examination of the patients will be used to evaluate the presence of apical lesion, size of the lesion, and PAI index. Microbiological examination (evaluation of UFC/ml) will be carried out to assess the disinfection of the root canals. The success rate of the treatment will also be assessed. Endodontic treatment will be carried out in accordance with habitual standards and practices. PDT will be applied with diode laser (660 nm, 100 mW) and methylene blue will be used as photosensitizer (PS). Patients of the Endodontics Service of Universidad San Sebastián (Santiago campus) will be recruited for the study.

DETAILED DESCRIPTION:
The object of the present study is to compare the effectiveness of conventional endodontic treatment with that of endodontic treatment combined with PDT in patients with apical lesion. A randomized, clinical, superiority trial will be carried out, controlled, blinded and masked, with 3 parallel arms.

The patient sample will be randomized in 3 treatment groups: the first is the placebo group which will receive conventional endodontic treatment (ET) and a simulated treatment with the equipment in which no radiation will be emitted; the second group will receive conventional ET associated with PDT with diode laser at 660 nm, fluence 10 s/canal; and the third group will receive conventional ET associated with PDAT with laser at 660 nm, 20 s/canal. The photosensitizer used in the PDT will be methylene blue.

Clinical and radiographic examination of all the patients will be used to obtain baseline values (T0) and values 6 months post-treatment (T1). The presence and size of apical lesion will be assessed at T0 and T1, the percentage reduction of the lesion will be calculated and the PAI index will be used as a scoring system to assess the lesion. The success rate will be assessed for each group 6 months after completion of the treatment. Disinfection of the root canals will be assessed by analysis of colony formation (ufc/ml); biological samples will be taken with paper cones inserted into the root canals to the apical region at two moments: Baseline (before treatment, T0); after instrumentation with PDT (experimental groups) and without PDT (placebo group). Adverse events will be analysed; a serious adverse event for this study is any unfavourable odontological event that the investigators believe to bear a causal relation with the experimental intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for this study must comply with the following for randomization:

1. Adult patients of either sex
2. No general biological risk
3. At least 1 molar with pulp necrosis and apical lesion

Exclusion Criteria:

1. Pregnancy
2. Patients requiring complex dental rehabilitation due to major coronal destruction
3. Individuals with cognitive disability making conventional treatment impossible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in lesion size. | From treatment at 6 months
  The lesion will be measured vertically and horizontally, and the size difference between the start of treatment and 6 months after treatment will be evaluated. The lesion will also be evaluated by the PAI index score. Interpretation of radiographs and PAI scores will be carried out by experienced endodontists.

SECONDARY OUTCOMES:
Disinfection of the root canals | before treatment (T0) and after treatment (T1)
  Disinfection of the root canals will be evaluated by analysis of colony formation (ufc/ml). To assess colony formation (ufc/ml) in the root canal, biological samples will be taken with paper cones inserted into the root canals to the apical region at two moments: Baseline (before treatment, T0); after instrumentation with PDT (experimental groups) and without PDT (placebo group). Three paper cones will be inserted into the root canals for 30 s. Routine microbiological analysis will be performed. Disinfection of the canal will be evaluated by comparing colony formation in each group at T0 and T1. Which treatment promotes the greatest disinfection will also be determined.
Success rate | From treatment at 6 months
  Success rate of the treatment, measured after 6 months, based on the clinical results (absence of clinical signs and symptoms) and on the radiographic results (diminution of the lesion and absence of root resorption, PAI index score). The analyses will be carried out by two calibrated researchers, who will be blinded to the patient's assignment to a treatment group. The success rate will be assessed for each group 6 months after completion of ET.

OTHER OUTCOMES:
adverse events | From treatment at 6 months
  Primary inferential analysis will be based on intention to treat. A protocol will be used to analyse the result variable 'adverse effects' to avoid underestimation of its magnitude. All adverse events will be recorded that occur from entry into the study until completion of treatment. A serious adverse event for this study is any unfavourable odontological event that the investigators believe to bear a causal relation with the experimental intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nilton Alves, PhD, Principal Investigator — Universidad de La Frontera
Locations (1):
- Universidad San Sebastián, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alves N, Deana NF, Abarca J, Monardes H, Betancourt P, Zaror C. Root Canal Disinfection in Permanent Molars with Apical Lesion by Antimicrobial Photodynamic Therapy: Protocol for a Blind Randomized Clinical Trial. Photobiomodul Photomed Laser Surg. 2024 May;42(5):366-374. doi: 10.1089/photob.2023.0186. PMID 38776543